CLINICAL TRIAL: NCT05344521
Title: A Phase I, Single-blind, Randomized Study of the Safety and Efficacy of Cellularized Integra® Using Autologous Burn-derived Stem Cells
Acronym: Integra®-SC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: AFP Innovation Fund (Other); Ontario Institute for Regenerative Medicine (Unknown); Stem Cell Network (Other)
Responsible Party: Principal Investigator, Marc Jeschke, Vice President of Research, Medical Director Burn Unit, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15229
Record Dates: First submitted 2022-03-24; First posted 2022-04-25 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Burns
Keywords: Stem Cells; Wound Healing; Cicatrix; Skin, Artificial
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Intervention Model Description: Integra®-SC will be applied to one area of the body and acellular Integra® will be applied to another. Determination of the location of the Integra® control or Integra®-SC application will be assigned using simple randomization. The wound areas will be appropriately matched for body surface area and depth of the wound.
Who Masked: Participant
Masking Description: This is a single-blind study where the participant will not know which area is covered with Integra®-SC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): After removal of the temporary wound coverage (allograft), Integra® is applied directly onto the wound surface.
  Interventions: Device: Integra®
- Integra®-SC (Experimental): After removal of the temporary wound coverage (allograft), Integra®-SC is applied to the contralateral area of the site where Integra® is applied.
  Interventions: Device: Integra®-SC

INTERVENTIONS:
Device: Integra® — A commercially available dermal bovine matrix that is widely used for wound and burn care, Integra® Dermal Regeneration Template licensed device (Medical Device Active License Listing No. 229).
  Arms: Control
Device: Integra®-SC — A combination of Integra® incorporated with 5,000-20,000 cells/cm2 of autologous burned derived stem cells.
  Arms: Integra®-SC

SUMMARY:
Burn injuries are one of the most severe skin injuries and lead to a complex wound healing response. When the skin is wounded, stem cells in the skin must respond fast to help repair the injured tissue. The damaged skin of burn patients contains cells that are still alive and have typical stem cell characteristics. Because stem cells are so important for wound healing, the investigators have combined them with an existing skin substitute, Integra®, to examine the potential wound healing benefits of these stem cells. This is an investigational treatment and a first in-human trial. The purpose of this study is to test the safety of using a patient's own stem cells combined with Integra®, which the investigators call Integra®-Stem Cells (Integra®-SC). The investigators hypothesize that Integra®-SC will result in improved wound healing, better scar quality, and decreased scar formation at one-year post-injury.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years.
* Total body surface area (TBSA) ≥ 5%.
* Full-thickness burn requiring operative procedures.
* Admitted ≤ 120 hours following burn.
* Injury location includes a contralateral area.

Exclusion Criteria:

All participants meeting any of the following exclusion criteria at baseline will be excluded from participation in this study:

* Patients who are moribund.
* Known infection with any of the following: Human Immunodeficiency Virus (HIV), Hepatitis B, Hepatitis C, Human T-lymphotropic Virus (HTLV), Syphilis, or West Nile Virus.
* Injury location limited to face and/or hands.
* Pregnancy.
* Active cancer and currently undergoing treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety - Number of participants with surgical site infections | Acute hospitalization (1-4 months post admission depending on severity of injury)
  The primary outcome of this study is safety. In order to assess the safety of Integra®-SC, surgical site infections that require an additional (unplanned) operation will be recorded as an in-hospital complication.
Safety - Number of participants with non-healing wounds | Acute hospitalization (1-4 months post admission depending on severity of injury)
  The primary outcome of this study is safety. In order to assess the safety of Integra®-SC, non-healing wounds that require an additional (unplanned) operation will be recorded as an in-hospital complication.
Safety - Number of patients with poor scarring requiring additional (unplanned) operation | Discharge to to 1 year post-discharge
  The primary outcome of this study is safety. In order to assess the safety of Integra®-SC, poor scarring requiring an additional (unplanned) operation will be recorded as a late-onset complication.

SECONDARY OUTCOMES:
Time of wound healing | Acute hospitalization (1-4 months post admission depending on severity of injury)
  Time from wound excision to 95% healing of the burned area will be recorded. Photography and evaluation of wounds will occur at enrollment, operation days, dressing take-downs, and discharge from hospital.
Quality of skin regeneration - Arterial bleeding from the wound site | Acute hospitalization (1-4 months post admission depending on severity of injury)
  Arterial bleeding from the wound site will be recorded to assess the quality of skin regeneration. Photography and evaluation of wounds will occur at enrollment, operation days, dressing take-downs, and discharge from hospital.
Quality of skin regeneration - Signs of wound infection | Acute hospitalization (1-4 months post admission depending on severity of injury)
  Classic signs of wound infection will be recorded to assess the quality of skin regeneration. Photography and evaluation of wounds will occur at enrollment, operation days, dressing take-downs, and discharge from hospital.
Quality of skin regeneration - Detachment of Integra®-SC | Acute hospitalization (1-4 months post admission depending on severity of injury)
  The detachment of the entire Integra®-SC from the wound site will be recorded to assess the quality of skin regeneration. Photography and evaluation of wounds will occur at enrollment, operation days, dressing take-downs, and discharge from hospital.
Quality of skin regeneration - Abnormal scar formation | Acute hospitalization (1-4 months post admission depending on severity of injury)
  The formation of hypertrophic scars or keloids will be recorded to assess the quality of skin regeneration. Photography and evaluation of wounds will occur at enrollment, operation days, dressing take-downs, and discharge from hospital.
Scar Formation - Vascularity of the healed area | Discharge to 1 year post-discharge
  Vascularity of the healed area is assessed as part of the Vancouver Scar Scale to evaluate scar formation over time. Vascularity is scored from 0 to 3, with higher scores indicating worse outcomes. Photography and evaluation of treated area for scar formation will be assessed at outpatient follow-ups at approximately 30 days, 60 days, 90 days, 180 days, and 365 days post-discharge (with 2-4 weeks deviation). Follow-ups typically take place in-person at clinic visits, but may take place online via a secure platform.
Scar formation - Pigmentation of the healed area | Discharge to 1 year post-discharge
  Pigmentation of the healed area is assessed as part of the Vancouver Scar Scale to evaluate scar formation over time. Pigmentation is scored from 0 to 2, with higher scores indicating worse outcomes. Photography and evaluation of treated area for scar formation will be assessed at outpatient follow-ups at approximately 30 days, 60 days, 90 days, 180 days, and 365 days post-discharge (with 2-4 weeks deviation). Follow-ups typically take place in-person at clinic visits, but may take place online via a secure platform.
Scar formation - Pliability of the healed area | Discharge to 1 year post-discharge
  Pliability of the healed area is assessed as part of the Vancouver Scar Scale to evaluate scar formation over time. Pliability is scored from 0 to 5, with higher scores indicating worse outcomes. Photography and evaluation of treated area for scar formation will be assessed at outpatient follow-ups at approximately 30 days, 60 days, 90 days, 180 days, and 365 days post-discharge (with 2-4 weeks deviation). Follow-ups typically take place in-person at clinic visits, but may take place online via a secure platform.
Scar formation - Height of the healed area | Discharge to 1 year post-discharge
  The height of the healed area is assessed as part of the Vancouver Scar Scale to evaluate scar formation over time. Height is scored from 0 to 3, with higher scores indicating worse outcomes. Photography and evaluation of treated area for scar formation will be assessed at outpatient follow-ups at approximately 30 days, 60 days, 90 days, 180 days, and 365 days post-discharge (with 2-4 weeks deviation). Follow-ups typically take place in-person at clinic visits, but may take place online via a secure platform.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Jeschke, MD PhD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada